CLINICAL TRIAL: NCT01376531
Title: Influence of Continuous Veno-venous Hemodialysis on Cerebrovascular Autoregulation in Patients With Acute Renal Failure
Brief Title: Influence Continuous Veno-venous Hemodialysis the Autoregulation
Acronym: dARICUCVVH
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Patrick Schramm, Senior Physician, Johannes Gutenberg University Mainz
Other Study IDs: 837.041.10 2
Record Dates: First submitted 2011-06-15; First posted 2011-06-20 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Acute Renal Failure
Keywords: acute renal failure; cerebrovascular autoregulation; transcranial Doppler; continuous veno-venous hemodialysis
MeSH Terms: conditions — Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute renal failure: patients at intensive care unit with definition of acute renal failure and the need for continuous veno-venous hemodialysis
  Interventions: Procedure: continuous veno-venous hemodialysis

INTERVENTIONS:
Procedure: continuous veno-venous hemodialysis — continuous veno-venous hemodialysis
  Other Names: CVVHD

SUMMARY:
The aim of the study is to characterize the influence of continuous veno-venous hemodialysis on the cerebrovascular autoregulation.

DETAILED DESCRIPTION:
Patients at the intensive care unit who suffered acute renal failure with the need of continuous veno-venous hemodialysis will be investigated with continuous veno-venous hemodialysis and in a time window without continuous veno-venous hemodialysis to investigate the influence of continuous veno-venous hemodialysis on the cerebrovascular autoregulation.

ELIGIBILITY:
Inclusion Criteria:

* acute renal failure
* need for continuous veno-venous hemodialysis
* age >18 Years

Exclusion Criteria:

* Sepsis
* Preexisting cerebral illness
* traumatic brain injury
* Meningitis or encephalitis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at ICU with acute renal failure and the need of continuos veno-venous hemodialysis
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline cerebrovascular autoregulation to cerebrovascular autoregulation during continuous veno-venous hemodialysis | 1 Year
  Is there an influence of continuous veno-venous hemodialysis at the cerebrovascular autoregulation, which would be a side effect with limiting use in patients with brain injury or the need of intensive monitoring of cerebral perfusion pressure in this patients.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schramm, MD, Principal Investigator — Department of Anesthesiology, University medicine Mainz, Germany
Locations (1):
- University medical centre, Mainz, Germany

REFERENCES:
- [Result] Schramm P, Closhen D, Wojciechowski J, Berres M, Klein KU, Bodenstein M, Werner C, Engelhard K. Cerebrovascular autoregulation in critically ill patients during continuous hemodialysis. Can J Anaesth. 2013 Jun;60(6):564-9. doi: 10.1007/s12630-013-9912-z. Epub 2013 Mar 28. PMID 23536386